CLINICAL TRIAL: NCT02691000
Title: The Light Heart Study: Daily Light Box Use for Depressive Symptoms in Patients With Stage B Heart Failure
Acronym: Light-Heart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Retirement Research Foundation (Other)
Responsible Party: Principal Investigator, Jeanne Maglione, Assistant Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 151558
Record Dates: First submitted 2016-01-29; First posted 2016-02-24 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Depression; Stage B Heart Failure
Keywords: depression; depressive symptoms; stage b heart failure; bright white light; light therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright White Light (BWL) Litebook (Experimental): Participants will be instructed to use the BWL Litebook for an hour every day for 8 weeks.
  Interventions: Device: LiteBook
- Dim Red Light (DRL) Litebook (Placebo Comparator): Participants will be instructed to use the DRL (comparison condition) Litebook for an hour every day for 8 weeks.
  Interventions: Device: LiteBook

INTERVENTIONS:
Device: LiteBook — Light therapy using a Bright White Light Litebook for 1 hour each morning for 8 weeks. This is the experimental intervention.
  Arms: Bright White Light (BWL) Litebook
Device: LiteBook — Light therapy using a Dim Red Light Litebook for 1 hour each morning for 8 weeks. This is the control.
  Arms: Dim Red Light (DRL) Litebook

SUMMARY:
The Light-Heart study is a randomized, double-blind, controlled trial investigating the effects of bright white light (BWL) therapy on depressive symptoms, quality of life, and functioning in patients with Stage B heart failure. The study is a randomized, double-blind, controlled trial of 8 weeks of morning BWL therapy compared with morning dim red light (DRL) treatment in older (60 years or older) 122 Stage B (early, asymptomatic) HF patients.

DETAILED DESCRIPTION:
The Light-Heart study is randomized, double-blind, controlled trial of 8 weeks of morning BWL therapy, compared with DRL in older, Stage B HF patients with clinically significant levels of depressive symptoms. The primary hypothesis of the proposed study is that compared to DRL, BWL therapy will be associated with a significantly greater reduction in depressive symptoms. Important information about compliance and tolerability associated with the BWL intervention in Stage B HF patients will also be gathered. The investigators will examine whether BWL therapy is associated with greater improvements in quality of life and subjective functioning compared to DRL. Finally, the researchers will investigate whether BWL is associated with a sustained improvement in depressive symptoms 2 and 4 weeks following the end of the intervention compared to DRL.

One hundred twenty-two older adults (≥60 years) with Stage B HF and depressive symptoms (Beck Depression Inventory/BDI score ≥10) will be recruited from several University of California, San Diego (UCSD) and Veteran's Affairs (VA) cardiology clinics. The baseline assessment will include evaluation of depressive symptoms (BDI), quality of life (Quality of Life Enjoyment and Satisfaction questionnaire), subjective functioning (Short Form-36), and an assessment of patient expectations regarding the study intervention (single question, 5 point scale). These measures will be assessed again after 4 and 8 weeks of treatment and at 2 and 4 weeks following the end of the BWL therapy intervention along with side effects (Frequency, Intensity, and Burden of Side Effects Rating).

Participants will be randomized to receive BWL (n=61) or DRL (n=61) light therapy boxes (Litebook® Elite; Litebook® Inc., Medicine Hat, CA) to use at home for 60 minutes each morning for 8 weeks. If participants are currently receiving treatment (e.g. antidepressant therapy), participants will continue their usual treatment while in the study. Participants will be told that the effects of a particular light therapy protocol on mood and functioning is being investigated. Participants will be made aware that there is a treatment condition of interest and a comparison condition and that participants will be randomly assigned to one or the other group. Participants will not be told that different colors of light are being used or that BWL is the treatment of interest. The Litebooks® will look identical except for the color of the light. Weekly telephone calls will encourage compliance, and compliance meters will record when the Litebooks® are turned on or off. A blood sample will also be collected from each patient to assess for biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years
* Written informed consent
* BDI score ≥ 10
* Stage B heart failure diagnosis
* no antidepressant pharmacotherapy or on stable dose of antidepressant (>8 weeks)
* on stable dose of cardiac medications (>8 weeks)

Exclusion Criteria:

* self-reported history of bipolar disorder
* psychiatric diagnoses by Structured Clinical Interview for the Diagnostic and Statistical Manual (DSM) (ie; bipolar disorder, schizophrenia, schizoaffective disorder, major neurocognitive disorder)
* serious suicide or homicide risk (outpatient care judged unsafe)
* recent initiation or change of dose in antidepressant or cardiac medications (within past 8 weeks)
* current use of supplements with putative effects on mood or sleep (e.g St. John's Wort, melatonin)
* recent initiation of evidence based psychotherapy for mood
* prior use of BWL therapy
* unstable medical illness requiring hospitalization
* uncontrolled seizure disorder
* retinopathies
* macular degeneration
* shift work

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms will be assessed with the Beck Depression Inventory. | baseline and at 8 week

SECONDARY OUTCOMES:
The Short Form (SF)-36 questionnaire will be used to assess QOL and subjective functioning. | Baseline and at 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Maglione, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient information will remain confidential.

REFERENCES:
- [Background] Abramson J, Berger A, Krumholz HM, Vaccarino V. Depression and risk of heart failure among older persons with isolated systolic hypertension. Arch Intern Med. 2001 Jul 23;161(14):1725-30. doi: 10.1001/archinte.161.14.1725. PMID 11485505
- [Background] Ahmedani BK, Solberg LI, Copeland LA, Fang-Hollingsworth Y, Stewart C, Hu J, Nerenz DR, Williams LK, Cassidy-Bushrow AE, Waxmonsky J, Lu CY, Waitzfelder BE, Owen-Smith AA, Coleman KJ, Lynch FL, Ahmed AT, Beck A, Rossom RC, Simon GE. Psychiatric comorbidity and 30-day readmissions after hospitalization for heart failure, AMI, and pneumonia. Psychiatr Serv. 2015 Feb 1;66(2):134-40. doi: 10.1176/appi.ps.201300518. Epub 2014 Nov 1. PMID 25642610
- [Background] Cameron IM, Reid IC, MacGillivray SA. Efficacy and tolerability of antidepressants for sub-threshold depression and for mild major depressive disorder. J Affect Disord. 2014 Sep;166:48-58. doi: 10.1016/j.jad.2014.04.078. Epub 2014 May 9. PMID 25012410
- [Background] Desan PH, Weinstein AJ, Michalak EE, Tam EM, Meesters Y, Ruiter MJ, Horn E, Telner J, Iskandar H, Boivin DB, Lam RW. A controlled trial of the Litebook light-emitting diode (LED) light therapy device for treatment of Seasonal Affective Disorder (SAD). BMC Psychiatry. 2007 Aug 7;7:38. doi: 10.1186/1471-244X-7-38. PMID 17683643
- [Background] Frasure-Smith N, Lesperance F. Depression--a cardiac risk factor in search of a treatment. JAMA. 2003 Jun 18;289(23):3171-3. doi: 10.1001/jama.289.23.3171. No abstract available. PMID 12813125
- [Background] Jiang W, Alexander J, Christopher E, Kuchibhatla M, Gaulden LH, Cuffe MS, Blazing MA, Davenport C, Califf RM, Krishnan RR, O'Connor CM. Relationship of depression to increased risk of mortality and rehospitalization in patients with congestive heart failure. Arch Intern Med. 2001 Aug 13-27;161(15):1849-56. doi: 10.1001/archinte.161.15.1849. PMID 11493126
- [Background] Jimenez JA, Mills PJ. Neuroimmune mechanisms of depression in heart failure. Methods Mol Biol. 2012;934:165-82. doi: 10.1007/978-1-62703-071-7_9. PMID 22933146
- [Background] Leppamaki SJ, Partonen TT, Hurme J, Haukka JK, Lonnqvist JK. Randomized trial of the efficacy of bright-light exposure and aerobic exercise on depressive symptoms and serum lipids. J Clin Psychiatry. 2002 Apr;63(4):316-21. PMID 12000205
- [Background] Lieverse R, Van Someren EJ, Nielen MM, Uitdehaag BM, Smit JH, Hoogendijk WJ. Bright light treatment in elderly patients with nonseasonal major depressive disorder: a randomized placebo-controlled trial. Arch Gen Psychiatry. 2011 Jan;68(1):61-70. doi: 10.1001/archgenpsychiatry.2010.183. PMID 21199966
- [Background] Loving RT, Kripke DF, Elliott JA, Knickerbocker NC, Grandner MA. Bright light treatment of depression for older adults [ISRCTN55452501]. BMC Psychiatry. 2005 Nov 9;5:41. doi: 10.1186/1471-244X-5-41. PMID 16283925
- [Background] Naus T, Burger A, Malkoc A, Molendijk M, Haffmans J. Is there a difference in clinical efficacy of bright light therapy for different types of depression? A pilot study. J Affect Disord. 2013 Dec;151(3):1135-7. doi: 10.1016/j.jad.2013.07.017. Epub 2013 Aug 7. PMID 23972661
- [Background] Rutledge T, Reis VA, Linke SE, Greenberg BH, Mills PJ. Depression in heart failure a meta-analytic review of prevalence, intervention effects, and associations with clinical outcomes. J Am Coll Cardiol. 2006 Oct 17;48(8):1527-37. doi: 10.1016/j.jacc.2006.06.055. Epub 2006 Sep 26. PMID 17045884
- [Background] Terman M, Terman JS. Light therapy for seasonal and nonseasonal depression: efficacy, protocol, safety, and side effects. CNS Spectr. 2005 Aug;10(8):647-63; quiz 672. doi: 10.1017/s1092852900019611. PMID 16041296
- [Background] Tuunainen A, Kripke DF, Endo T. Light therapy for non-seasonal depression. Cochrane Database Syst Rev. 2004;2004(2):CD004050. doi: 10.1002/14651858.CD004050.pub2. PMID 15106233